CLINICAL TRIAL: NCT04044612
Title: Effect of Knee Bracing on Improving Pain & Disability, Physical Performance, Physical Activity and Femoral Cartilage Deformation in Individuals With Medial Compartment Knee Osteoarthritis
Brief Title: Effect of Knee Bracing on Improving Pain & Disability
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: American Orthotic and Prosthetic Association (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 18-2363
Record Dates: First submitted 2019-08-01; First posted 2019-08-05 (Actual); Last update posted 2021-03-08 (Actual); Status verified 2021-03

CONDITIONS: Knee Osteoarthritis
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Medial Unloader Brace (Experimental)
  Interventions: Other: Medial Unloader Brace

INTERVENTIONS:
Other: Medial Unloader Brace — medial knee unloader braces use a three point bending system to increase space in the medial tibiofemoral compartment during weight bearing

SUMMARY:
The overall purpose of the proposed pilot study is to establish the feasibility of conducting a clinical trial by evaluating the preliminary effects of 8 weeks of knee bracing on physiological measures of self-reported pain and disability, physical performance, physical activity, as well as femoral cartilage deformation in individuals with medial compartment knee osteoarthritis (OA). The investigators will recruit 36 symptomatic knee OA patients for the pilot study. The investigators will evaluate a class of braces (two different models will be used) designed to correct genu varum. The purpose of the study is to evaluate changes in these novel outcomes following the use of a class of braces used to reduce medial tibiofemoral compartment compression used for 8 weeks. This pilot study will inform a larger future trial to determine the efficacy of bracing on decreasing disability and disease progression in patients with knee osteoarthritis.

ELIGIBILITY:
Inclusion Criteria:

Participants must:

* have a physician diagnosis of knee OA in the medial compartment and exhibit symptomatic knee OA, which the investigators will define as a normalized, person based, Western Ontario and McMaster Universities Arthritis Index (WOMAC) function subscale score > 31 (out of 100 points, indicating most dysfunction).
* have had a knee radiograph taken within the previous 6 months.
* be between the ages of 40 and 75 years old will be included.

Exclusion Criteria:

Participants will be excluded if they have:

* been diagnosed with a cardiovascular condition restricting exercise;
* had a corticosteroid or hyaluronic acid injection in the involved knee in the previous 2 weeks;
* a pacemaker;
* a neurodegenerative condition;
* rheumatoid arthritis;
* cancer;
* neural sensory dysfunction over the knee;
* a BMI over 35;
* history of lower extremity orthopaedic surgery in the past year;
* a history of a traumatic knee injury in the past 6 months;
* any history of a total knee arthroplasty in either extremity; or
* a diagnosed, non-reconstructed knee ligament tear.
* the need of an assistive device to walk.

The investigators will also exclude pregnant women, as well as women who are trying to get pregnant or plan to get pregnant during the study.

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2018-12-01 (Actual); Primary Completion 2020-03-31 (Actual); Study Completion 2020-03-31 (Actual)

PRIMARY OUTCOMES:
Percentage Change in WOMAC Function score from Baseline to 8 weeks | Baseline, Week 8 (Followup)
  The Western Ontario and McMasters Osteoarthritis Index (WOMAC) is a self-reported measure of disability. The physical function consists of 17 items and asks about the magnitude of difficulty when ascending and descending stairs, rising from sitting, standing, bending, walking, getting in/out of a car, shopping, putting on and taking off socks, rising from bed, lying in bed, getting in and out of the bath, sitting, getting on and off the toilet, completing heavy household duties, and completing light household duties. Each item is presented in a 5 point Likert-type format and uses the following descriptors for possible answer choices none, mild moderate, severe, and extreme. Each descriptor corresponds to an ordinal scale of 0-4. The scores are summed for the items in each subscale, with a total possible range from 0-68. Higher scores indicate greater amounts of functional limitations.
Percentage Change in Physical Activity Scale for the Elderly from Baseline to 8 weeks | Baseline, Week 8 (Followup)
  Physical Activity Scale for the Elderly (PASE) scores are calculated from weights and frequency values for each of 12 types of activity. Responses to the first question about sitting activities are not scored. The scale is continuous with higher scores indicating greater physical activity
Percentage Change in 30-s chair-stand test from Baseline to 8 weeks | Baseline, Week 8 (Followup)
  The number of times that an individual can sit and stand in 30 seconds.
Percentage Change in 20 meter fast-paced walk test from Baseline to 8 weeks | Baseline, Week 8 (Followup)
  The investigators will time the amount of seconds it takes to walk 20 meters.
Percentage Change in Stair-climb test from Baseline to 8 weeks | Baseline, Week 8 (Followup)
  The investigators will time the amount of seconds it takes to walk up and down a flight of stairs.
Percentage Change in Femoral Cartilage Cross-sectional area from Baseline to 8 weeks | Baseline, Week 8 (Followup)
  The investigators will measure the amount of cartilage cross-sectional area on the anterior femur before and after 3000 steps of walking. A greater change in cross-sectional area is determined to be more more cartilage deformation.

CONTACTS AND LOCATIONS:
Overall Officials: Brian Pietrosimone, Principal Investigator — University of North Carolina, Chapel Hill
Locations (1):
- Motion Science Institute, Chapel Hill, North Carolina, United States

IPD SHARING:
Plan to Share IPD: Yes
Deidentified individual data that supports the results will be shared beginning 9 to 36 months following publication provided the investigator who proposes to use the data has approval from an Institutional Review Board (IRB), Independent Ethics Committee (IEC), or Research Ethics Board (REB), as applicable, and executes a data use/sharing agreement with UNC
Time Frame: 9 to 36 months following publication
Access Criteria: Investigator who proposes to use the data has IRB, IEC, or REB approval and executed a data use/sharing agreement with UNC.